CLINICAL TRIAL: NCT07185126
Title: Developing Innovative PTSD Treatment for Children: Reconsolidation of Traumatic Memories Protocol™ for Children (RTM-C Protocol)
Brief Title: Developing Innovative PTSD Treatment for Children
Acronym: ChildrenRTM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Viktoriia Gorbunova (Other)
Collaborators: Charitable Foundation Voices of Children (Unknown); Quresta, Inc. (Unknown)
Responsible Party: Sponsor-Investigator, Viktoriia Gorbunova, Vice President, Global Institute for Mental Health Innovations, Networking and Development a.s.b.l.
Organization: Global Institute for Mental Health Innovations, Networking and Development a.s.b.l. (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: № 07062025
Record Dates: First submitted 2025-08-25; First posted 2025-09-22 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Post Traumatic Stress Disorder PTSD
Keywords: RTM; Reconsolidation of Traumatic Memories; PTSD; Post Traumatic Stress Disorder; Children
MeSH Terms: conditions — Combat Disorders; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: This is a non-randomized, single-arm interventional pilot study. All participants will receive the RTM-C Protocol. Following the parent session (for consent and orientation), children will complete six structured RTM-C Protocol sessions, followed by diagnostic assessments at 1 and 6 months. This pilot study uses an open-label design with no masking, as the intervention requires active therapist and child engagement. The primary purpose is treatment: to test whether the RTM-C Protocol reduces post-traumatic stress symptoms and improves child functioning, while also assessing feasibility and acceptability among children, parents, and providers.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Reconsolidation of traumatic memories in Children (RTM-C) (Experimental): Experimental: RTM-C Protocol. All participants will receive the RTM-C Protocol intervention, an adapted version of the adult RTM Protocol™ designed for children aged 6-14 with post-traumatic stress symptoms. Parents and children complete follow-up assessments at 1 and 6 months to measure outcomes.
  Interventions: Behavioral: Reconsolidation of traumatic memories

INTERVENTIONS:
Behavioral: Reconsolidation of traumatic memories — The intervention begins with a parent session to review history, provide orientation, and obtain consent. Each child then attends six individual therapy sessions with a trained RTM specialist. Sessions use imagination exercises, "film-like" replay of traumatic memories in modified formats (e.g., black-and-white, fast-forward, backwards), and structured state-interruption techniques to reduce fear and distress. Animated instructions and cardboard "cinema" and "skreen" models may be used to support comprehension if needed.

SUMMARY:
This study is testing a new version of a treatment called the Reconsolidation of Traumatic Memories Protocol for Children (RTM-C Protocol). The RTM Protocol™ is already proven to help adults with post-traumatic stress disorder (PTSD) by reducing distressing memories, flashbacks, and nightmares. The children's version is specially adapted to meet the needs of children aged 6-14, using child-friendly language, games, and animated tools.

The purpose of this study is to find out whether the RTM-C Protocol can safely and effectively reduce post-traumatic stress symptoms in children who have experienced trauma. We also want to know whether children, parents, and therapists find the method acceptable and easy to use.

Children and their parents will take part in a series of sessions with a trained specialist. Parents will join an initial session to provide information and give consent. Children will then have up to six therapy sessions, during which they learn to safely "replay" their difficult memories in imaginative ways that reduce their fear. Parents and children will complete questionnaires about symptoms before and after the sessions, as well as at 1 and 6 months after completion.

Study Question: Can the RTM-C Protocol reduce post-traumatic stress symptoms in children and improve their daily functioning (such as relationships, learning, and happiness)?

Study Hypothesis: RTM-C Protocol will lead to a significant reduction in PTSD symptoms in children, with improvements maintained at follow-up, and will be rated as acceptable and feasible by children, parents, and therapists.

DETAILED DESCRIPTION:
Post-traumatic stress disorder (PTSD) in children is a serious mental health problem that can develop after exposure to traumatic events such as war, violence, displacement, accidents, loss of loved ones, or abuse. PTSD in children is associated with intrusive memories, nightmares, physiological hyperarousal, avoidance of reminders, irritability, concentration difficulties, and impairments in family life, schooling, and social relationships. Although evidence-based psychological treatments exist for adults, there remains a major gap in effective, developmentally appropriate, and scalable interventions for children.

The Reconsolidation of Traumatic Memories (RTM) Protocol™ is a brief, non-pharmacological intervention originally developed for adults with PTSD. It is based on cognitive and neurobiological models of memory reconsolidation and dissociation. The RTM Protocol™ uses imagery to help individuals safely reprocess traumatic memories through a series of dissociative and imaginative steps (e.g., replaying memories in black-and-white, running them backwards, speeding them up). This process reconsolidates the traumatic memory in a less distressing form, leading to a rapid reduction in flashbacks, nightmares, and distress responses. The RTM Protocol™ in adults has demonstrated strong clinical effectiveness across several clinical trials, with high acceptability and minimal risk of re-traumatisation.

The children's version of the RTM Protocol™ (RTM-C Protocol) retains the essential procedural components of the adult method but is carefully adapted to meet developmental needs. Adaptations include:

* Child-friendly language and explanations.
* The use of play-based and imaginative exercises.
* Animated instructional videos and a cardboard "cinema" and "skreen" models to guide children through visualisation steps.
* Additional therapist strategies for emotional support, grounding, and engagement.
* Structured parental involvement before, during and after treatment sessions.

RTM-C Protocol™ is designed to reduce post-traumatic symptoms without requiring children to recount painful details. It is therefore less burdensome and carries minimal risk of retraumatisation compared with traditional trauma-focused exposure therapies.

Study design and stages. This pilot study involves a mixed-methods evaluation. A single-arm pilot with approximately 40-48 children, each treated by one of 20-24 trained RTM Protocol specialists. Children will complete six RTM-C Protocol sessions (plus parental sessions and diagnostic follow-ups). Outcomes will be measured at baseline, post-treatment, 1 month, and 6 months after treatment. Qualitative feedback will also be collected from specialists through structured focus groups.

Intervention procedures. RTM-C Protocol involves six structured sessions with the child, preceded by a parent session and followed by diagnostic follow-ups (at 1 month and 6 months after treatment), with both children and parents, to assess sustained outcomes.

Each session lasts approximately 60 minutes and follows a detailed, structured protocol. Animated instructions and cardboard "cinema" and "skreen" models are used as supportive tools only when verbal instructions are insufficient. Therapists are trained to avoid unnecessary use of tools that could prolong the session or burden the child. Children are rewarded at the end of sessions with small positive reinforcements (stickers, drawings, short games) to enhance engagement.

Therapist training and fidelity. All providers are certified RTM specialists. They receive additional one-day training in the RTM-C Protocol. Fidelity is supported through the use of protocol texts, animations, and visual tools, and monitored by session checklists and coaching. Feedback from therapists on usability, language, and feasibility will be used to refine the protocol before larger rollout.

Safety considerations. The RTM-C Protocol emphasises "stress-free recall." Children are not asked to provide detailed verbal descriptions of traumatic events. The therapist interrupts immediately if distress arises and redirects the child's focus to a safe, neutral task. Work with traumatic material proceeds only once the child has demonstrated the ability to switch states reliably during practice (clear disengagement from imagery, reorientation to the present, ability to make eye contact, relaxed affect). These safeguards minimise the risk of re-traumatisation.

Data collection and measures. The study uses the CATS-2 (Child and Adolescent Trauma Screen) as the primary outcome measure, administered to both children and parents. The CATS-2 provides scores for PTSD symptoms and functional impairment in relationships, learning, leisure, and happiness. Additional brief questionnaires and structured interviews will assess acceptability and feasibility from both families and providers. Data will be collected at baseline, post-treatment, and at 1- and 6-month follow-ups.

Data protection. All identifying information is anonymised using codes. Personal data are securely stored in locked cabinets and password-protected computers in Ukraine. Anonymised datasets may be transferred via secure, certified platforms. Only trained RTM specialists have access to identified data. Researchers analyse only anonymised data.

Scientific hypothesis. The study hypothesises that the RTM-C Protocol will significantly reduce PTSD symptoms in children, with effects maintained at 1- and 6-month follow-ups, and that children, parents, and therapists will find the intervention safe, acceptable, and feasible.

Significance. If effective, the RTM-C Protocol will provide an innovative, scalable, and low-burden treatment for PTSD in children. It could address a major unmet need in child mental health, particularly in humanitarian and post-conflict contexts. The pilot study in Ukraine is a first step toward larger implementation and evaluation, and findings will contribute to global knowledge on child-appropriate trauma interventions.

ELIGIBILITY:
Inclusion Criteria:

* Age 6-14 years at enrolment.
* PTSD symptoms present: CATS-2 (Parent) total ≥15 at screening.
* Functional impact: impairment endorsed in ≥1 CATS-2 domain (relationships, leisure, learning, happiness).
* Consent/assent: written parent/guardian consent and child assent obtained.
* Availability: child and caregiver can attend parent session + 6 treatment sessions and complete 1- and 6-month follow-ups.
* Language/comprehension: child can understand session instructions and participate in tasks (with supports as needed).
* Therapist check of readiness: during Session 1 practice, child demonstrates reliable break state (disengages from imagery, re-orients to present, maintains eye contact, relaxed affect).

Exclusion Criteria:

* Acute comorbid mental disorder.
* Concurrent trauma-focused psychotherapy planned or ongoing during the study period.
* Inability to understand/follow instructions due to cognitive impairment or other reasons that preclude participation.
* Medical/neurological condition or situational factors (e.g., inability to commit to visits) that, in the investigator's judgment, would make participation unsafe or compromise study integrity.

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2025-09-20 (Actual); Primary Completion 2026-02-20 (Estimated); Study Completion 2026-08-20 (Estimated)

PRIMARY OUTCOMES:
Change in post-traumatic stress symptoms (CATS-2 total score) | Baseline (pre-intervention, Session 1), 1-month follow-up, and 6-month follow-up.
  The primary outcome is the change in total PTSD symptom severity, measured by the Child and Adolescent Trauma Screen - 2 (CATS-2). Both child self-report and parent-report versions will be administered. The CATS-2 assesses frequency of PTSD symptoms such as intrusive memories, nightmares, hyperarousal, avoidance, and negative thoughts/emotions. The CATS-2 is a validated screening and outcome tool for children and adolescents exposed to trauma. Change in CATS-2 total score reflects clinical improvement in PTSD symptoms and is the most direct measure of RTM-C effectiveness.

CONTACTS AND LOCATIONS:
Overall Officials: Viktoriia Gorbunova, ScD, Principal Investigator — Global Institute for Mental Health Innovations, Networking and Development
Locations (1):
- Charitable Foundation Voices of Children, Kyiv, Ukraine

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared outside the therapists who will collect data. This decision is based on the high sensitivity of the data, which involves trauma histories and mental health information from children. Even with de-identification, the small sample size and the vulnerability of the population create a risk of re-identification. For these reasons, only anonymised data will be shared with researchers, and only aggregated results will be shared through publications and presentations.

REFERENCES:
- [Result] Astill Wright L, Horstmann L, Holmes EA, Bisson JI. Consolidation/reconsolidation therapies for the prevention and treatment of PTSD and re-experiencing: a systematic review and meta-analysis. Transl Psychiatry. 2021 Sep 3;11(1):453. doi: 10.1038/s41398-021-01570-w. PMID 34480016
- [Result] Sturt J, Rogers R, Armour C, Cameron D, De Rijk L, Fiorentino F, Forbes T, Glen C, Grealish A, Kreft J, Meye de Souza I, Spikol E, Tzouvara V, Greenberg N. Reconsolidation of traumatic memories protocol compared to trauma-focussed cognitive behaviour therapy for post-traumatic stress disorder in UK military veterans: a randomised controlled feasibility trial. Pilot Feasibility Stud. 2023 Oct 13;9(1):175. doi: 10.1186/s40814-023-01396-x. PMID 37833734
- [Result] Gorbunova V, Hampton R. The Reconsolidation of Traumatic Memories Protocol's adjustments to the remote treatment of injured Ukrainian military personnel in hospital settings. Eur J Psychotraumatol. 2025 Dec;16(1):2499410. doi: 10.1080/20008066.2025.2499410. Epub 2025 May 19. PMID 40387497
- See also: GlobalinMind Announcement of the Project — https://www.globalinmind.eu/portfolio-collections/our-project/developing-innovative-ptsd-treatment-for-children
- See also: Voices of Children Announcement of the Project — https://voices.org.ua/en/news/v-ukrayini-vpershe-stvoryuyut-dityachu-versiyu-innovacijnogo-metodu-roboti-z-travmoyu

DOCUMENTS (3):
  • Study Protocol (2025-11-18): https://cdn.clinicaltrials.gov/large-docs/26/NCT07185126/Prot_003.pdf
  • Informed Consent Form: Parent Consent Form (2025-11-18): https://cdn.clinicaltrials.gov/large-docs/26/NCT07185126/ICF_004.pdf
  • Informed Consent Form: Child Assent Form (2025-11-18): https://cdn.clinicaltrials.gov/large-docs/26/NCT07185126/ICF_005.pdf